CLINICAL TRIAL: NCT02268292
Title: The Effects of Home Bicycle Exercise Program on Hyperlipidemia, Hypertension, Blood Sugar Control, Muscle Strength and Aerobic Capacity
Brief Title: Home Bicycle Exercise and Aerobic Capacity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, Taichung Veterans General Hospital, Taichung Veterans General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG12147
Record Dates: First submitted 2014-09-27; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Metabolic Cardiovascular Syndrome
Keywords: Metabolic syndrome; Diabetes; Muscle strength; Aerobic exercise; Bicycle; Brain-derived neurotrophic factor
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bicycle Exercise (Experimental): Bicycle Exercise for 12 weeks
  Interventions: Behavioral: bicycle exercise

INTERVENTIONS:
Behavioral: bicycle exercise — All enrolled subjects received a scheduled twelve-week exercise program. A commercially available bicycle (Giant CS800, Taichung, Taiwan) with an indoor bicycle stand (Giant Cyclotron Mag, Taichung, Taiwan) was used as the home exercise training modality.

SUMMARY:
The subjects with MetS or type 2 diabetes were enrolled for this exercise-training program. All participators underwent an indoor bicycle exercise for twelve weeks. In addition to demographic data and biochemical tests were determined after an overnight fasting. Extension of muscle strength was detected in the dominant lower extremity.

DETAILED DESCRIPTION:
This prospective open-labeled study was conducted in Taichung Veterans General Hospital. The adult participants with metabolic syndrome and/or type 2 diabetes were enrolled. MetS. The procedures were fully explained to all subjects before the cardiopulmonary exercise test. ll enrolled subjects received a scheduled twelve-week program for exercise-training program. A commercially available bicycle with an indoor bicycle trainer are used as the home exercise training modality. All medications were not allowed to be changed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult with metabolic syndrome or type 2 diabetes

Exclusion Criteria:

* hyperglycemic crisis or HbA1c > 12%;
* serum creatinine levels greater than 200 mmol/L;
* acute or chronic infectious diseases;
* limitations in the ability to undertake regular exercise

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome | 12 weeks
  Components of metabolic syndrome based on the modified Third Report of the National Cholesterol Education Program (NCEP) criteria

SECONDARY OUTCOMES:
Muscle strength | 12 weeks
  A Biodex Isokinetic Dynamometer (Biodex Medical Systems, Inc., Shirley, New York, USA) was used to evaluate the muscle strength of the subjects
Brain-derived neurotrophic factor | 12 weeks
  Serum concentration of Brain-derived neurotrophic factor (enzyme immunoassay method, R&D Systems, Minneapolis, U.S.A.)
Arterial stiffness | 12 weeks
  Pulse wave velocity

REFERENCES:
- [Derived] Tsai SW, Chan YC, Liang F, Hsu CY, Lee IT. Brain-derived neurotrophic factor correlated with muscle strength in subjects undergoing stationary bicycle exercise training. J Diabetes Complications. 2015 Apr;29(3):367-71. doi: 10.1016/j.jdiacomp.2015.01.014. Epub 2015 Feb 7. PMID 25682570